CLINICAL TRIAL: NCT05581056
Title: Evaluation of the Evolution of Quality of Life in Relation to Naso-sinus Symptomatology Under Treatment With CFTR Modulators in Children Aged 6 to 11 Years With Cystic Fibrosis With Compatible Mutation
Brief Title: Evaluation of the Evolution of Quality of Life in Relation to Naso-sinus Symptomatology Under Treatment With CFTE Modulators in Children Aged 6 to 11 Years With Cystic Fibrosis With Compatible Mutation
Acronym: MUCOSINTRIO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0836
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Naso sinusal symptoms
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CFTR modulators group: Children between 6 and 11 years old that will be treated by CFTR modulators.
  Interventions: Drug: CFTR modulators

INTERVENTIONS:
Drug: CFTR modulators — Introduction of CFTR modulators by pneumologists for pneumologic issues

SUMMARY:
Cystic fibrosis is a multi-organ disease. It most often results from a genetic mutation, the delta F508 mutation, which prevents the expression of the CFTR 'régulateur de conductance transmembranaire de la fibrose kystique) protein. If the poor prognosis of the disease is correlated to the pulmonary damage, we observe, at the naso-sinus level, a significant functional impact, with chronic rhino-sinusal damage that can alter the quality of life of patients. In addition to this functional impact, some studies suggest that these chronic naso-sinus attacks are involved in the creation of a bacterial reservoir that is secondarily responsible for pulmonary colonization and therefore partly responsible for the poor prognosis of the disease.

The clinical and paraclinical examinations can be used to determine the extent of these disorders. Their functional impact can be assessed using quality of life questionnaires such as the SN-5 scale.

Treatment with CFTR modulators in patients with mutations compatible with the treatment seems to transform their vital prognosis. The scientific rationale of this treatment consists in restoring the activity of the CFTR protein, allowing the recovery of the hydro-electrolytic balance of the mucous secretions, and thus reducing the viscosity of the biological fluids. The various studies carried out all prove a dramatic improvement in pulmonary parameters under treatment, with very limited toxicity.

A marketing authorization for this treatment has been issued on the European market for patients over 18 years of age in 2020, for children over 12 years of age in 2021, and will soon be issued for children aged between 6 and 11 years.

Since the pathophysiology of pulmonary and nasosinus involvement are similar, and since this treatment will be marketed for children between 6 and 11 years of age, we expect an improvement in rhino-sinus symptomatology. To date, clinical studies have focused primarily on pulmonary outcomes. There are only few publications dealing with the evolution of nasosinus symptomatology under treatment, and none concerning the pediatric population.

The aim of our study is to evaluate the evolution of naso-sinusal symptomatology under treatment with CFTR modulators in children aged 6 to 11 years. This will allow us to confirm or deny the interest of these treatments in the extra-pulmonary manifestations of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 11 years of age
* Compatible genotype and patient treated with KAFTRIO (treatment initiation is independent of this study)

Exclusion Criteria:

* Refusal of the child or the holder of parental authority to participate in the study.
* Child not affiliated to a social security system and under legal protection
* Holder of parental authority who does not master the French language

Secondary Exclusion Criteria:

* Sinus surgery during the observation period
* Poor tolerance of the treatment (pneumological opinion)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 6 and 11 years of age
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Evolution of quality of life, evaluated with SN-5 scale. | Baseline, 6 months, 12 months
  The analysis of the primary endpoint is based on the analysis of a quantitative variable, the mean SN-5 score of the entire population, before and at one year after treatment.
  This statistical analysis is based on a comparison of two averages: the average SN-5 score before treatment and the average SN-5 score at one year after treatment in 90 patients.
  In previous studies, after external validation, a change of at least 0.57 points in the SN-5 score is used as a threshold to consider at least a slight clinical change

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petit G, Coudert A, Hermann R, Truy E, Bonjour M, Reix P, Ayari S. Effects of Elexacaftor-Tezacaftor-Ivacaftor on Nasal and Sinus Symptoms in Children With Cystic Fibrosis. Pediatr Pulmonol. 2025 Jan;60(1):e27493. doi: 10.1002/ppul.27493. PMID 39868969